CLINICAL TRIAL: NCT00003693
Title: Phase I Study of Dolastatin-10 in Acute Leukemias, Myelodysplastic Syndromes and Chronic Myeloid Leukemia in Blast Phase
Brief Title: Dolastatin 10 in Treating Patients With Refractory or Relapsed Acute Leukemia, Myelodysplastic Syndrome, or Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM98-187; U01CA062461 (NIH); P30CA016672 (NIH); MDA-DM-98187 (Other: UT MD Anderson Cancer Center); NCI-T98-0001; CDR0000066796 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-03-23 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; previously treated myelodysplastic syndromes; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Blast Crisis; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic | interventions — dolastatin 10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MTD Group (Experimental)
  Interventions: Drug: Dolastatin 10

INTERVENTIONS:
Drug: Dolastatin 10 — IV bolus once every 3 weeks.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of dolastatin 10 in treating patients who have refractory or relapsed acute leukemia, chronic myelogenous leukemia in blast phase, or myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose and dose limiting toxicity of dolastatin 10 in patients with chronic myelogenous leukemia in blast phase, refractory or relapsed acute leukemia, or myelodysplastic syndromes. II. Assess the possible antileukemia effect of this treatment in these patients.

OUTLINE: This is a dose escalation study. Patients receive dolastatin 10 intravenous (IV) bolus once every 3 weeks. Patients receive 2-12 courses of therapy in the absence of disease progression and unacceptable toxicity. In the absence of dose limiting toxicity (DLT) in the first cohort of 3 patients, subsequent cohorts of 3 patients each receive escalating doses of dolastatin 10. If DLT occurs in 2 of 3 patients at a given dose level, then dose escalation ceases and the next lower dose is declared the maximum tolerated dose. Patients are followed until death.

PROJECTED ACCRUAL: This study will accrue up to 25 patients within 8 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically diagnosed chronic myelogenous leukemia in blastic phase, refractory or relapsed acute leukemia, or myelodysplastic syndromes (refractory anemia with excess blasts (RAEB), RAEB in transformation, or chronic myelomonocytic leukemia)

PATIENT CHARACTERISTICS: Age: Not specified Performance status: 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin no greater than 1.5 mg/dL SGPT no greater than 2 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance greater than 60 mL/min Other: Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since prior chemotherapy and recovered (unless evidence of rapid disease progression) Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 1998-12-18 (Actual); Primary Completion 2001-10-30 (Actual); Study Completion 2001-10-30 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Dolastatin | Assessed with each 3 week cycle
  Maximum tolerated dose defined by dose limiting toxicity of dolastatin.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org